CLINICAL TRIAL: NCT07139561
Title: Oral Health in Hands: A Digital Intervention to Improve Oral Health Practices in Children
Brief Title: A Digital Intervention to Improve Oral Health Practices
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Arshed Muhammad, PhD, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: BMU-BBC
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Digital Intervention; Oral Health Behavior Change
MeSH Terms: interventions — Oral Health

STUDY DESIGN:
Intervention Model Description: It is two arm randomized control trial
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Investigators and outcome assessors will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will be given no intervention other than they will receive routinely
- Intervention arm (Experimental): Oral Health in Hands - Parent Digital Program: The intervention includes daily reminders with two brushing cues and one snack tip to reinforce habits. Weekly quizzes with 3-5 questions assess knowledge, while photo/video tasks such as "Show your foam smile" or "Healthy lunchbox challenge" keep engagement high. Gamification features badges for streaks like a 7-day brushing badge or snack swap champion. Parents track brushing, flossing, and snack swaps via a 1-tap tracker, supported by an optional moderated WhatsApp group.
  Interventions: Behavioral: Oral Health in Hands - Parent Digital Program

INTERVENTIONS:
Behavioral: Oral Health in Hands - Parent Digital Program — The 16-week parent-focused digital intervention aims to improve oral health practices in children aged 6-10 by empowering parents through structured, engaging, and cost-effective activities. Parents receive daily reminders, including two brushing cues and one snack tip, to reinforce healthy routines. Weekly quizzes with 3-5 questions enhance knowledge retention, while interactive photo or video tasks such as "Show your foam smile" or "Healthy lunchbox challenge" promote family involvement and fun. Gamification strategies include awarding digital badges for streaks, such as the 7-day brushing badge and snack swap champion, to maintain motivation. Parents track brushing, flossing, and snack swaps using a simple 1-tap tracker, ensuring easy and consistent reporting. An optional moderated WhatsApp group provides a platform for sharing tips, photos, and encouragement, fostering a supportive peer community. The intervention combines education, habit formation, and social support to sustainab
  Arms: Intervention arm

SUMMARY:
This study evaluates a 16-week parent-focused digital intervention to improve oral health practices in children aged 6-10 through daily reminders, quizzes, challenges, gamification, and behavior tracking, supported by an optional moderated WhatsApp group for peer engagement and motivation.

DETAILED DESCRIPTION:
The intervention includes daily reminders with two brushing cues and one snack tip to reinforce habits. Weekly quizzes with 3-5 questions assess knowledge, while photo/video tasks such as "Show your foam smile" or "Healthy lunchbox challenge" keep engagement high. Gamification features badges for streaks like a 7-day brushing badge or snack swap champion. Parents track brushing, flossing, and snack swaps via a 1-tap tracker, supported by an optional moderated WhatsApp group.

ELIGIBILITY:
Inclusion Criteria:

* Parents or primary caregivers of children aged 6-10 years.
* Child must be free from major systemic illnesses or developmental disabilities that could interfere with oral hygiene practices.
* Parent/caregiver owns a smartphone with access to WhatsApp or similar digital platform.
* Ability to read or understand Urdu or English instructions.
* Willingness to participate for the full 12-week duration and provide informed consent.

Exclusion Criteria:

* Children with serious medical conditions (e.g., immunodeficiency, congenital anomalies) that may affect oral health.
* Parents or children currently enrolled in another oral health education or digital intervention program.
* Children who have received professional oral health education or structured interventions within the past 4 months.
* Parents/caregivers unwilling or unable to comply with digital reporting and participation requirements.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Estimated)
Dates: Start 2025-08-18 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-18 (Estimated)

PRIMARY OUTCOMES:
Oral health practices | 4-months
  Oral health practices by using the WHO Child Oral Health Questionnaire: o assess children's oral health practices through a structured set of questions. These questionnaires typically cover knowledge, attitude, and practices related to oral hygiene, including frequency of brushing, use of fluoride toothpaste, and dental visits. The score is used to evaluate the overall oral health practices of the child, often categorized as good, fair, or poor.
Oral Hygiene | 4-months
  Oral Hygiene will be assessed by the presence of debris (plaque) and calculus (tartar) on selected tooth surfaces, measured by the Simplified Oral Hygiene Index (OHI-S) Individual Debris Index (DI-S) and Calculus Index (CI-S): Each of the six surfaces is scored individually for both debris and calculus using a 0-3 scale: 0: No debris or calculus is present. 1: Debris or calculus covers less than one-third of the surface. 2: Debris or calculus covers between one-third and two-thirds of the surface. 3: Debris or calculus covers more than two-thirds of the surface. Good: 0.0 - 1.2 Fair: 1.3 - 3.0 Poor: 3.1 - 6.0

SECONDARY OUTCOMES:
Plaque score | 4-months
  Oral Hygiene will be assessed by the presence of debris (plaque) and calculus (tartar) on selected tooth surfaces, measured by the Simplified Oral Hygiene Index (OHI-S) Individual Debris Index (DI-S) and Calculus Index (CI-S): Each of the six surfaces is scored individually for both debris and calculus using a 0-3 scale: 0: No debris or calculus is present. 1: Debris or calculus covers less than one-third of the surface. 2: Debris or calculus covers between one-third and two-thirds of the surface. 3: Debris or calculus covers more than two-thirds of the surface. Good: 0.0 - 1.2 Fair: 1.3 - 3.0 Poor: 3.1 - 6.0
Gingival score | 4-months
  Gingival score assessed by the gingival score index: 0: Normal gingiva, no inflammation. 1: Mild inflammation - slight color change and edema (swelling), no bleeding on probing. 2: Moderate inflammation - redness, edema, glazing, and bleeding on probing. 3: Severe inflammation - marked redness, edema, ulceration, and tendency towards spontaneous bleeding. The index typically uses a scale of 0 to 3, with 0 representing normal gingiva and higher scores indicating increasing severity of inflammation

CONTACTS AND LOCATIONS:
Locations (4):
- Pakistan (4):
  - White house grammar School, Chak Number Two North Branch, Punjab Province
  - Baqai Medical complex school, Karachi, Sindh
  - Saleem ullah fahmi memorial school unit 1, Karachi, Sindh
  - Saleem ullah fahmi school baqai Medical complex gharo, Karachi, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No
Only the study protocol, statistical plan, and results will be shared in publications in peer-reviewed journals

REFERENCES:
- [Background] Li X, Xu ZR, Tang N, Ye C, Zhu XL, Zhou T, Zhao ZH. Effect of intervention using a messaging app on compliance and duration of treatment in orthodontic patients. Clin Oral Investig. 2016 Nov;20(8):1849-1859. doi: 10.1007/s00784-015-1662-6. Epub 2015 Dec 2. PMID 26631059
- [Background] Lee JA, Choi M, Lee SA, Jiang N. Effective behavioral intervention strategies using mobile health applications for chronic disease management: a systematic review. BMC Med Inform Decis Mak. 2018 Feb 20;18(1):12. doi: 10.1186/s12911-018-0591-0. PMID 29458358
- [Background] Machado RA, de Souza NL, Oliveira RM, Martelli Junior H, Bonan PRF. Social media and telemedicine for oral diagnosis and counselling in the COVID-19 era. Oral Oncol. 2020 Jun;105:104685. doi: 10.1016/j.oraloncology.2020.104685. Epub 2020 Apr 10. No abstract available. PMID 32291154
- [Background] Abduljalil HS, Abuaffan AH. 'Knowledge and practice of mothers in relation to dental health of pre-school children. Adv Genet Eng. 2016;5:1-7. https://doi.org/10.4172/2169-0111.1000153.
- [Background] Alqarni AA, Alfaifi HM, Aseeri NA, Gadah T, Togoo RA. Efficacy of a Self-Designed Mobile Application to Improve Child Dental Health Knowledge among Parents. J Int Soc Prev Community Dent. 2018 Sep-Oct;8(5):424-430. doi: 10.4103/jispcd.JISPCD_195_18. Epub 2018 Oct 8. PMID 30430070